CLINICAL TRIAL: NCT05998395
Title: Single Patient Study of JAK/STAT Inhibition in CNS Kohlmeier-Degos Disease
Brief Title: JAK/STAT Inhibition in CNS Kohlmeier-Degos Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001517; 001517-H
Record Dates: First submitted 2023-08-17; First posted 2023-08-21 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Kohlmeier Degos Disease With Neurologic Involvement; Kohlmeier-Degos Disease
Keywords: Rare Small Vessel Vasculopathy Of Unknown Etiology; Kohlmeier Degos Disease With Neurologic Involvement; Interferon Related Disease
MeSH Terms: conditions — Malignant Atrophic Papulosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib in Participants with CNS Kohlmeier-Degos Disease (Experimental): Ruxolitinib at 5 mg twice a day (BID) for 1 week and then at 10 mg BID for 13-73 weeks and 1 week of 5 mg BID before stopping ruxolitinib.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib at 5 mg twice a day (BID) for 1 week and then at 10 mg BID for 13-73 weeks and 1 week of 5 mg BID before stopping ruxolitinib.
  Other Names: Jakafi

SUMMARY:
Background:

Kohlmeier-Degos (K-D) is a rare disease that leads to the inflammation and/or blockage of small blood vessels in many organs; these can include the skin, eyes (rare), small bowels, lungs, heart, and the brain and spinal cord (central nervous system, or CNS). There are no known effective treatments for K-D that affects the CNS.

Objective:

To test a drug (ruxolitinib) in a person with K-D affecting the CNS.

Eligibility:

This study is designed to treat 1 adult participant with K-D affecting the CNS.

Design:

The participant will be screened:

They will have a physical exam and blood tests.

They will have skin biopsies: Small samples of skin will be removed.

They will have a lumbar puncture: A needle will be inserted in his back to draw fluid from the space around the spinal cord.

They will have a magnetic resonance imaging (MRI) scan: they will lie on a table that slides into a tube to take pictures of their brain and spinal cord.

They will see a doctor who specializes in nerves.

Ruxolitinib is a tablet taken by mouth. The participant will take the drug twice a day for up to 26 weeks. The dosage may change over time.

The participant will have up to 7 clinic visits in 28 weeks. Each visit will be 1 to 3 days. MRI scans, biopsies, lumbar punctures, and other blood tests will be repeated on different visits. The participant may receive follow-up phone calls between visits. The participant will report any adverse effects. Unscheduled visits may be needed if new symptoms develop.

The last follow-up will be 4 weeks after the last dose of the study drug.

DETAILED DESCRIPTION:
Study Description:

This single patient protocol will provide off-label treatment with a JAK/STAT ( Janus kinases/ Signal transducer and Activator of Transcription proteins) inhibitor to a patient with Kohlmeier Degos disease (K-D) with neurologic involvement. We hypothesize that ruxolitinib, which targets type I IFN (Interferons ) and IFN-gamma signaling, will attenuate various neurological manifestations of K-D that are observed clinically, radiologically or in abnormal laboratory findings in our K-D patient. This will help reduce IFN signaling in a manner that may slow or halt the disease progression as measured by the endpoints established below.

Objectives:

Primary Objective:

To test the hypothesis that JAK/STAT inhibition by ruxolitinib will delay progression of neuroradiological manifestations of our one patient with neurological involvement of K-D disease.

Exploratory Objectives:

1. Assess changes in immune cell proportion using single cell RNAseq (scRNA-seq) in biospecimens such as skin, cerebrospinal fluid (CSF) and blood after 13 weeks and up to 73 weeks of ruxolitinib treatment.
2. Assess changes in plasma/serum cytokines levels and IFN scores as well as biomarker assays in CSF/ blood samples after 13 weeks and up to 73 weeks of ruxolitinib treatment..
3. To test the hypothesis that ruxolitinib will stabilize or improve clinical neurologic exams in this patient.

Endpoints:

Primary Endpoint:

The primary endpoint is stability or regression of existing enhancing lesions or no development of new enhancing lesions in the brain and spine observed in MRI evaluation after 13 weeks and up to 73 weeks of ruloxitinib (10 mg BID) compared to pre-treatment MRI images.

Exploratory endpoints of this study are clinical and potential surrogate biomarker efficacy data, including:

1. Changes in transcriptome/RNA expression determined by scRNA-seq in skin, CSF and peripheral blood mononuclear cells (PBMCs) between baseline measurements and after 13 weeks and up to 73 weeks of treatment.
2. Attenuation of plasma/serum cytokine levels and IFN scores as well as biomarker assays in CSF and blood samples between the baseline visit and after 13 weeks and up to 73 weeks of treatment.
3. Stability OR improvement of motor and/or sensory function on clinical neurologic exams between the baseline visit and after 13 weeks and up to 73 weeks of treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study design was constructed to treat one participant with CNS Kohlmeier Degos Disease. Therefore, there are no specific inclusion criteria.

EXCLUSION CRITERIA:

* Active life-threatening infections
* Hemoglobin <7 g/dL
* Platelet counts < 50 K /mcL
* Neutropenia (ANC <0.5 x k/mcL)
* Lymphopenia (ALC <0.2 x k/mcL)
* LFTs (liver function test) > 3 x time upper limit
* eGFR/CreatCr < 30 mL/min

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia D Cudrici, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant results data will be made available 6 months after publication date for a period of 5 year by sending a request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available 6 months after publication date for a period of 5 year.
Access Criteria: send request to cornelia.cudrici@nih.gov

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001517-H.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable or no Lesions Developed Based on MRI Neurological Involvement of K-D Disease Following Ruloxitinib
Description: The primary endpoint is stability or regression of existing enhancing lesions or no development of new enhancing lesions in the brain and spine observed in MRI evaluation after 13 weeks and up to 73 weeks of ruloxitinib (10 mg BID) compared to pre-treatment MRI images.
Time Frame: Baseline, up to 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease
Number analyzed (Participants) | 1
Participants
  Stabilization of Lesions | 1
  Regression of Lesions | 0
  New Lesions | 0

2. Primary Outcome: Number of Participants With Stable or no Lesions Developed Based on MRI Neurological Involvement of K-D Disease Following Ruloxitinib
Description: as for outcome 1
Time Frame: 13 weeks up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease
Number analyzed (Participants) | 1
Participants
  Stabilization of Lesions | 0
  Regression of Lesions | 0
  New Lesions | 1

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Arm/Group | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease (N=1)
Worsening Sacral wound abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib in Participants With CNS Kohlmeier-Degos Disease (N=1)
Depression (Psychiatric disorders) | 1 (1)
Abnormal MRI (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT05998395/Prot_SAP_001.pdf
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05998395/ICF_000.pdf